CLINICAL TRIAL: NCT04824417
Title: A Randomized Controlled Trial to Compare the Clinical Outcomes With Six Months of Therapy With Oral Itraconazole Versus Oral Voriconazole for Management of Treatment naïve Subjects With Chronic Pulmonary Aspergillosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGI/IEC/2019/002366
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pulmonary Aspergillosis
Keywords: cpa; aspergillosis
MeSH Terms: conditions — Aphakia, congenital primary; Aspergillosis | interventions — Itraconazole; Voriconazole

STUDY DESIGN:
Intervention Model Description: Randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Oral itraconazole
  Interventions: Drug: Itraconazole 200 mg
- Intervention (Experimental): Oral voriconazole
  Interventions: Drug: Voriconazole 200mg

INTERVENTIONS:
Drug: Itraconazole 200 mg — Control
  Arms: Control
Drug: Voriconazole 200mg — Comparator
  Arms: Intervention

SUMMARY:
The current initial therapy for CPA is with six months of oral itraconazole. However, the response with six months of therapy has a response rate of 65-70% and has a relapse rate after stopping treatment of up to 50%. Voriconazole is a third-generation azole and a theoretical advantage of lower MICs compared to itraconazole. Also, oral voriconazole has good availability (95%) in fasting state. This is likely to improve the response rate and reduce the chances of relapse of chronic pulmonary aspergillosis. There is no head to head comparison of oral itraconazole with oral voriconazole. In this study we intent to compare the clinical outcomes with six months of therapy with oral itraconazole versus oral voriconazole for management of treatment naïve subjects with chronic pulmonary aspergillosis

DETAILED DESCRIPTION:
Aspergillus is a saprophytic fungus which is present normally in our surroundings and causes a large number of pulmonary diseases spreading through inhalational route. The spectrum of disease caused by aspergillus spp. is wide with the manifestations of the disease being governed primarily by the status of the underlying host immunity, which then determines the nature of the host-aspergillus interaction. Patients with an intact immunity have a more stable and indolent form of disease like aspergilloma whereas with a worsening immune status, the risk of invasive disease increases. Chronic pulmonary aspergillosis (CPA) and allergic bronchopulmonary aspergillosis (ABPA) are two of the commonest pulmonary manifestations seen in non-immunocompromised patients whereas invasive pulmonary aspergillosis being more common in the immunocompromised patients.(1-3) Estimates suggest that CPA affects around 3 million people across the globe, which may still be an under estimated number as the disease co exists with other pulmonary co-morbidities which make accurate diagnosis a pitfall. In India the annual incidence of CPA was estimated in 2011 and varied between 27,000-0.17 million cases, with different estimates. Based on the mortality rate for CPA which was estimated to be 15% annually, the 5-year prevalence of CPA was placed at 290,147 cases with 5-year prevalence rate being 24 per 100,000 in the same year.(4, 5) The disease confers significant morbidity and mortality, making it a significant burden for the society as well as the healthcare. Apart from the respiratory symptoms, CPA causes significant constitutional symptoms as well which adds to the misery of the patient. The diagnosis of CPA is based on presence of chronic symptoms, consistent radiology and demonstration of Aspergillus by direct (culture) or indirect (serological) methods.(1-3) Even though CPA is more of a disease spectrum but overall it is characterized by slowly progressive lung cavitation which may or may not show presence of mycetoma /fungal ball in patients with pre-existing structural lung diseases, even though other patterns have also been identified.

The treatment options majorly consist of medical management with at least 6-month long treatment with antifungal drugs - most significantly the azole groups. Itraconazole is the preferred azole for the treatment of CPA.(6-8) However the response with itraconazole is seen in around 60-75% of the subjects.(9) Moreover, about 30%-50% of the subjects have disease relapse that requires prolonged therapy. The lower response could be because of variable pharmacokinetics and drug absorption of oral itraconazole. Also, itraconazole has many drug interactions. Voriconazole is a third-generation azole and is currently the therapy of choice for invasive aspergillosis due to its lower minimal inhibitory concentration (MIC) values compared to itraconazole. In addition, the pharmacokinetics of voriconazole are not variable and oral form has a good bioavailability (up to 95%). In a previous study, the use of voriconazole resulted in radiological control in 97% of the subjects and a significant improvement in patients' symptoms but global success at six-months was only seen in 32% subjects.(10) However, despite being multicenter the study only included 48 subjects. Moreover, there was no control group and the authors did not use therapeutic dose monitoring. In addition, the study also included subjects with subacute invasive aspergillosis (SAIA). Thus, there is lack of information regarding the role of voriconazole in subjects with CPA. We hypothesize that the use of voriconazole will be associated with better treatment outcomes compared with oral itraconazole in treatment naïve subjects with CPA. In this randomized controlled trial, we compare the clinical outcomes of six months therapy with oral itraconazole with oral voriconazole in treatment naïve subjects with chronic pulmonary aspergillosis.

REFERENCES

1. Ullmann AJ, Aguado JM, Arikan-Akdagli S, Denning DW, Groll AH, Lagrou K, et al. Diagnosis and management of Aspergillus diseases: executive summary of the 2017 ESCMID-ECMM-ERS guideline. Clinical microbiology and infection : the official publication of the European Society of Clinical Microbiology and Infectious Diseases. 2018.
2. Patterson TF, Thompson GR, 3rd, Denning DW, Fishman JA, Hadley S, Herbrecht R, et al. Practice Guidelines for the Diagnosis and Management of Aspergillosis: 2016 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2016;63(4):e1-e60.
3. Denning DW, Cadranel J, Beigelman-Aubry C, Ader F, Chakrabarti A, Blot S, et al. Chronic pulmonary aspergillosis: rationale and clinical guidelines for diagnosis and management. The European respiratory journal. 2016;47(1):45-68.
4. Agarwal R, Denning DW, Chakrabarti A. Estimation of the burden of chronic and allergic pulmonary aspergillosis in India. PloS one. 2014;9(12):e114745.
5. Agarwal R. Burden and distinctive character of allergic bronchopulmonary aspergillosis in India. Mycopathologia. 2014;178(5-6):447-56.
6. Agarwal R, Aggarwal AN, Sehgal IS, Dhooria S, Behera D, Chakrabarti A. Performance of serum galactomannan in patients with allergic bronchopulmonary aspergillosis. Mycoses. 2015;58(7):408-12.
7. Agarwal R, Dua D, Choudhary H, Aggarwal AN, Sehgal IS, Dhooria S, et al. Role of Aspergillus fumigatus-specific IgG in diagnosis and monitoring treatment response in allergic bronchopulmonary aspergillosis. Mycoses. 2017;60(1):33-9.
8. Ashbee HR, Barnes RA, Johnson EM, Richardson MD, Gorton R, Hope WW. Therapeutic drug monitoring (TDM) of antifungal agents: guidelines from the British Society for Medical Mycology. J Antimicrob Chemother. 2014;69(5):1162-76.
9. Agarwal R, Vishwanath G, Aggarwal AN, Garg M, Gupta D, Chakrabarti A. Itraconazole in chronic cavitary pulmonary aspergillosis: a randomised controlled trial and systematic review of literature. Mycoses. 2013;56(5):559-70.
10. Cadranel J, Philippe B, Hennequin C, Bergeron A, Bergot E, Bourdin A, et al. Voriconazole for chronic pulmonary aspergillosis: a prospective multicenter trial. European journal of clinical microbiology & infectious diseases : official publication of the European Society of Clinical Microbiology. 2012;31(11):3231-9.

ELIGIBILITY:
Inclusion Criteria:

The cases will include treatment naïve consecutive subjects with chronic cavitary pulmonary aspergillosis (CPA). The diagnosis of CPA will be made by a multidisciplinary team (pulmonary physicians, radiologist and microbiologist) based on composite of clinical, radiological and microbiological criteria.(9, 10) This includes presence of all the following: (i) one or more clinical symptoms (persistent cough, recurrent hemoptysis, weight loss, malaise, fever and dyspnea) for ≥3 months; (ii) slowly progressive or persistent radiological findings (one or more cavities and surrounding fibrosis, infiltrates, consolidation, with or without fungal ball or progressive pleural thickening) on computed tomography (CT) of the thorax; (iii) immunological (A.fumigatus-specific IgG >27 mgA/L or positive Aspergillus precipitins) or microbiological evidence of Aspergillus infection (growth of Aspergillus in respiratory secretions or serum galactomannan index >0.6 or BALF galactomannan index >1.4); and, (iv) exclusion of other pulmonary disorders with similar presentation.

Exclusion Criteria:

Subjects with any of the following will be excluded: (i) failure to provide informed consent; (ii) patients on immunosuppressive drugs, intake of prednisolone (or equivalent) >10 mg for at least 3 weeks or a diagnosis of human immunodeficiency virus syndrome; (iii) intake antifungal azoles for >3 weeks in the preceding six months; (iv) subjects with active pulmonary infection due to mycobacterium tuberculosis or mycobacteria other than tuberculosis (MOTT); (v) subjects with others forms of pulmonary aspergillosis (allergic bronchopulmonary aspergillosis, chronic necrotizing aspergillosis and angio-invasive aspergillosis); and, (vi) pregnancy.

Ages: 13 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
proportion of subjects with an overall favourable response at the end of oral itraconazole therapy | six months

SECONDARY OUTCOMES:
number of relapses at six-months after completion of therapy | six months
adverse events due to itraconazole or voriconazole | six months

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Chest clinic, Chandigarh
  - Respiratory ICU, Department of Pulmonary Medicine, PGIMER, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sehgal IS, Agarwal R, Dhooria S, Prasad KT, Muthu V, Aggarwal AN, Rudramurthy SM, Garg M, Chakrabarti A. Oral itraconazole versus oral voriconazole for treatment-naive patients with chronic pulmonary aspergillosis in India (VICTOR-CPA trial): a single-centre, open-label, randomised, controlled, superiority trial. Lancet Infect Dis. 2025 Oct 29:S1473-3099(25)00537-7. doi: 10.1016/S1473-3099(25)00537-7. Online ahead of print. PMID 41175884